CLINICAL TRIAL: NCT04120857
Title: A Tele-Health Symptom Management Program for Patients With Heart Failure: Pall-Heart
Acronym: Pall-Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Jill Howie Esquivel, PhD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21320
Record Dates: First submitted 2019-09-24; First posted 2019-10-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
Keywords: stretching; exercise
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Control Group (No Intervention): Education provided for optional use
- Gentle Stretching and Education (Experimental): Gentle Stretching for 60 minutes twice weekly
  Interventions: Behavioral: Gentle Stretching

INTERVENTIONS:
Behavioral: Gentle Stretching — 60 minutes fo gentle stretching twice weekly for 8 weeks
  Other Names: Exercise
  Arms: Gentle Stretching and Education

SUMMARY:
Heart failure is common in adults and is the most common hospital diagnosis in older adults. Patients with heart failure suffer numerous distressing symptoms daily. Although palliative care can improve suffering, rural-dwelling heart failure patients have poor access to specialized palliative care. The investigators propose to pilot test a tele-health palliative care intervention, PALL-HEART, in rural dwelling heart failure patients who live in Virginia and Kentucky.

Study specific objectives are:

Primary Aims:

* AIM 1: Compare HF patients who participate in a home-delivered tablet-based HF health education and gentle stretching intervention, to a health education (HE) group on: a) HF symptoms (weight gain, breathlessness, fatigue), b) psychological symptoms (depression, diminished QOL, resilience, self-care, and heart rate variability), c) physical function (endurance, strength, balance), and d) health care utilization rates (ED visits, office visits, hospitalizations).
* Hypothesis 1: HF symptoms (weight gain, breathlessness, fatigue), psychological symptoms (depression, diminished QOL, resilience, self-care), physical function (endurance, strength, balance) will improve in the intervention group.
* Hypothesis 2: Health care utilization rates (ED visits, office visits, hospitalizations) will decrease in the intervention group.

Secondary:

* AIM 2: Acceptability - Acceptability of the intervention will be determined using: a) participation and satisfaction rates (participant logs), b) intervention retention rates, and c) barriers to participation (technology and participant motivation issues).
* Hypothesis: Subjects in the intervention group will have >80% participation and satisfaction rates and be willing to identify barriers to participation.

acceptability of the intervention for future refinement and large scale testing.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with reduced ejection fraction or Heart failure with preserved ejection fraction as seen by problem list in the EMR, is a patient in the heart failure clinic, or general cardiology clinic.
* ability to read, write and understand English;
* agree to participate and give informed consent;
* 19 years of age and older;
* telephone access;
* and NYHA class I-III with no changes in medications in 30 days (i.e. medical therapy is optimized).

Exclusion Criteria:

* are pregnant and/or breast feeding (self-reported)
* have a history of non-adherence with medications (as described by their provider or medical record);
* have had a hospitalization within the last 3 months for HF;
* have unstable angina; CABG, MI or biventricular pacemaker less than 6 weeks prior;
* have orthopedic impediments to stretching exercise;
* have severe COPD with a forced expiratory volume in one second less than 1 liter as measured by spirometry;
* have severe stenotic valvular disease;
* have a history of resuscitated sudden cardiac death without subsequent placement of an implantable cardioverter defibrillator;
* exercise more than 3 times weekly; currently engage in yoga at least 1 time per week;
* have cognitive impairment (as measured by the Mini-Cog)
* are living in a nursing home
* history of pulmonary arterial hypertension (PASP>60mmHg)
* other serious life-limiting co-morbidity, e.g. end stage cancer
* post-heart transplant (s/p OHT) or Left Ventricular Assist Device (LVAD)
* New York Heart Association Functional Class IV

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Heart Failure Somatic Perception Scale Questionnaire | 10 weeks
  This questionnaire measures symptoms of heart failure - The 18-item Somatic Perception Scale asks participants how much they are bothered by 18 symptoms of heart failure in the past week using 5 response options ranging from 0 (I did not have the symptom) to 5 (extremely bothersome). Scores are summed, with higher values indicating higher symptom burden. Scores range from 0-90 with higher values indicating higher symptom burden.
PROMIS questionnaire | 10 weeks
  This questionnaire screens for symptoms of depression. The 8-item questionnaire assesses self-reported negative mood (sadness, guilt), views of self (self- criticism, worthlessness), and social cognition (loneliness, interpersonal alienation) in the past week. The questionnaire uses 5 response options ranging from 0 (never) to 5 (always). Scores are summed, with higher values indicating higher risk for depression. The total raw score is converted into a T-score. The T-score rescales the raw score into a standardized score. The final score is a standardized score with a mean of 50 and a standard deviation of 10.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 10 weeks
  This questionnaire measures quality of life in people with heart failure. This questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. In the KCCQ, a summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Overall scores are transformed to a range of 0-100, in which higher scores reflect better health status. There are summary scores within the KCCQ and the overall summary score is created by the mean of Physical Limitation Score, Total Symptom Score, Quality of Life Score, and Social Limitation Score.
The Resilience Scale | 10 weeks
  The Resilience Scale is a 25-item administered questionnaire that measures an individual's ability to adapt over time to stressors in life. Scores on the summated scale range from 25 to 175, with higher scores indicating higher resilience. All of the items are positively worded. Items are measured on a 7-point scale from 1(strongly disagree) to 7 (strongly agree). Responses are summed to produce a total score where a higher score indicates higher resilience.
Self-Care for Heart Failure Index Questionnaire (SCHFI) | 10 weeks
  The Self-Care for Heart Failure Index Questionnaire (SCHFI) is a 39-item measure of heart failure self-care. The items range from never (1) to always (5). There are 3 subscales: maintenance scale, symptom perception, confidence scale, and management scale. All of the scales are scored in the same way and a total score is not computed. Separate scores for each scale are computed separately.
  In general, to standardize a scale score, 1) determine the maximum possible scale score, 2) subtract the number of items from the possible score, and 3) divide 100 by that result to identify a constant for that scale. To score the scale, sum item responses, subtract the number of items answered, and multiply by the constant.The higher the score, the greater the ability to care for heart failure symptoms within each subscale.
Endurance | 10 weeks
  2 step test - step alternating knees upward for 2 minutes
upper body strength - we will measure bicep strength by the number of hand weight lifts | 10 weeks
  participants are instructed to perform as many arm curls as possible for 30 seconds
lower body strength - we will measure quadricep strength by the number of times siting and standing in 30 seconds | 10 weeks
  participants are instructed to sit and then to stand as many times as possible in 30 seconds
balance | 10 weeks
  stand on 1 leg for as long as possible

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators who request the dataset. No individual personal or HIPPA identifiers will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: when data are analyzed and for 5 years.

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Ni H, Xu J. Recent Trends in Heart Failure-related Mortality: United States, 2000-2014. NCHS Data Brief. 2015 Dec;(231):1-8. PMID 26727546
- [Background] Zambroski CH, Moser DK, Bhat G, Ziegler C. Impact of symptom prevalence and symptom burden on quality of life in patients with heart failure. Eur J Cardiovasc Nurs. 2005 Sep;4(3):198-206. doi: 10.1016/j.ejcnurse.2005.03.010. PMID 15916924
- [Background] Rogers JG, Patel CB, Mentz RJ, Granger BB, Steinhauser KE, Fiuzat M, Adams PA, Speck A, Johnson KS, Krishnamoorthy A, Yang H, Anstrom KJ, Dodson GC, Taylor DH Jr, Kirchner JL, Mark DB, O'Connor CM, Tulsky JA. Palliative Care in Heart Failure: The PAL-HF Randomized, Controlled Clinical Trial. J Am Coll Cardiol. 2017 Jul 18;70(3):331-341. doi: 10.1016/j.jacc.2017.05.030. PMID 28705314
- [Background] Braun LT, Grady KL, Kutner JS, Adler E, Berlinger N, Boss R, Butler J, Enguidanos S, Friebert S, Gardner TJ, Higgins P, Holloway R, Konig M, Meier D, Morrissey MB, Quest TE, Wiegand DL, Coombs-Lee B, Fitchett G, Gupta C, Roach WH Jr; American Heart Association Advocacy Coordinating Committee. Palliative Care and Cardiovascular Disease and Stroke: A Policy Statement From the American Heart Association/American Stroke Association. Circulation. 2016 Sep 13;134(11):e198-225. doi: 10.1161/CIR.0000000000000438. Epub 2016 Aug 8. PMID 27503067
- [Background] Dracup K, Moser DK, Pelter MM, Nesbitt TS, Southard J, Paul SM, Robinson S, Cooper LS. Randomized, controlled trial to improve self-care in patients with heart failure living in rural areas. Circulation. 2014 Jul 15;130(3):256-64. doi: 10.1161/CIRCULATIONAHA.113.003542. Epub 2014 May 9. PMID 24815499
- [Background] Donesky D, Selman L, McDermott K, Citron T, Howie-Esquivel J. Evaluation of the Feasibility of a Home-Based TeleYoga Intervention in Participants with Both Chronic Obstructive Pulmonary Disease and Heart Failure. J Altern Complement Med. 2017 Sep;23(9):713-721. doi: 10.1089/acm.2015.0279. Epub 2017 Jun 27. PMID 28654302
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Pope C, Ziebland S, Mays N. Qualitative research in health care. Analysing qualitative data. BMJ. 2000 Jan 8;320(7227):114-6. doi: 10.1136/bmj.320.7227.114. No abstract available. PMID 10625273
- [Background] Martyn Hammersley. Challenging Relativism: The Problem of Assessment Criteria. Qual Inq. 2009 Jan 1;15(1):3-29.
- [Background] Clive Seale. Quality in Qualitative Research. Qual Inq. 1999 Dec 1;5(4):465-78